CLINICAL TRIAL: NCT05962242
Title: Circulating Tumor Modified HPV DNA-Guided Radiotherapy De-intensification of the Elective Neck (RaDEN) in Squamous Cell Carcinoma of the Head and Neck
Brief Title: HPV DNA-Guided Radiotherapy De-intensification of Head and Neck Squamous Cell Carcinoma
Acronym: HN001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christopher McLaughlin, MD, Assistant Professor of Radiation Oncology, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR220263
Record Dates: First submitted 2023-06-30; First posted 2023-07-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx
Keywords: Radiation Therapy; Radiotherapy; Head Cancer; Neck Cancer; Low Dose Radiation; HPV
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Participants on this study will undergo a reduced dose regimen starting with a boost to gross disease of 24 Gy, then 30-36 Gy to entire volume based on the plan for concurrent chemotherapy. Non-responders will receive a boost to the entire volume for an additional 10 Gy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reduce Dose without Concurrent Chemotherapy Non- Rapid Responder (Experimental): A reduced dose regimen of 24 Gy in 12 fractions to gross disease and intermediate nodes. Then 36 Gy in 18 fractions to entire volume. Non-responders will receive an additional boost of 10 Gy in 5 fractions to entire volume.
  Interventions: Radiation: Radiation Therapy
- Reduce Dose with Concurrent Chemotherapy Non-Rapid Responder (Experimental): A reduced dose regimen of 24 Gy in 12 fractions to gross disease and intermediate nodes. Then 30 Gy in 15 fractions to entire volume. Non-responders will receive an additional boost of 10 Gy in 5 fractions to entire volume.
  Interventions: Radiation: Radiation Therapy
- Reduce Dose without Concurrent Chemotherapy Rapid Responder (Experimental): A reduced dose regimen of 24 Gy in 12 fractions to gross disease and intermediate nodes. Then 36 Gy in 18 fractions to entire volume.
  Interventions: Radiation: Radiation Therapy
- Reduce Dose with Concurrent Chemotherapy Rapid Responder (Experimental): A reduced dose regimen of 24 Gy in 12 fractions to gross disease and intermediate nodes. Then 30 Gy in 15 fractions to entire volume.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — External Beam Radiation to Head and Neck

SUMMARY:
The study will evaluate the safety and effectiveness of a lower than standard dose of radiation for definitive or adjuvant treatment of head and neck squamous cell carcinomas.

DETAILED DESCRIPTION:
In squamous cell carcinomas of the head and neck, regional recurrence is rare within lymph node stations treated with elective radiation. However, radiotherapy to the neck is toxic, and leads to a variety of unpleasant side effects, especially coupled with concurrent systemic therapy. There is growing evidence from previous studies showing that lower radiation doses may be adequate in preventing locoregional recurrence of disease. The hypothesis is that lower dose of radiation will have equal effectiveness but less toxicity than standard approaches for the treatment of squamous cell carcinomas of the head and neck.

The study evaluates the effectiveness and safety of reduced dose radiotherapy for definitive and adjuvant treatment of Human papillomavirus (HPV) positive oropharyngeal squamous cell carcinomas.

Participants will be treated with a radiation therapy regimen that has a lower dose to less tissue area (dose and volume de-escalation) than standard of care radiation therapy. The dosing will be determined by whether concurrent chemotherapy will be given, results from on treatment HPV blood test called NavDx, physical exam, and imaging. On treatment NavDx results indicating a slow (non-rapid) response to the treatment will receive an additional boost of radiation. Routine NavDx testing will be performed to assess treatment response and recurrence. Participants will also be asked to complete surveys about overall health and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, ≥ 18 years of age
4. Pathologically proven diagnosis of squamous cell carcinoma of the oropharynx of any AJCC 8th edition stage.
5. Eligible for and planning to receive definitive treatment or adjuvant treatment with radiotherapy.
6. Participants who are receiving concurrent systemic anticancer therapy (e.g. chemotherapy or immunotherapy) for oropharyngeal cancer are eligible.

   1. For participants with T1-2 and N0 disease, chemotherapy is not required for eligibility. Participants may or may not receive chemotherapy per physician discretion.
   2. For participants with T3-4 and/or N+ disease, chemotherapy is required for eligibility.
7. Participants may receive investigational agents with prior approval from the Principal Investigator.
8. ECOG Performance Status of 0-2.
9. p16 positive HPV as determined by NavDx and immunohistochemistry
10. For females of reproductive potential: agreement to use adequate contraception during radiation treatment and for 6 months (or more if applicable based on other medications) after the end of radiation treatment.

Exclusion Criteria:

1. Evidence of distant metastatic disease
2. Prior history of radiotherapy to the head and/or neck
3. Had surgery for oropharyngeal cancer within 8 months of enrollment unless it was an incomplete oncologic surgery. Participant is eligible if the gross tumor was not completely removed.
4. Diagnosis of T3-4 and/or N+ disease with no plans to receive concurrent chemotherapy.
5. Diagnosis of a current or prior invasive malignancy (except non-melanoma skin cancer) unless the participant has been disease free for at least 3 years.
6. Participant is a prisoner
7. Known contraindications to head and neck radiation therapy such as ataxia telangiectasia or scleroderma.
8. Pregnancy or lactation
9. Active or severe co-morbidities as defined by the following:

   1. Unstable angina and/or congestive heart failure requiring hospitalization up to 180 days before registration
   2. Transmural myocardial infarction up to 180 days before registration
   3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   5. Hepatic insufficiency as determined by the treating clinician resulting in clinical jaundice and/or coagulation effects or severe liver dysfunction.
   6. Acquired immune deficiency syndrome (AIDS) based upon current CDC definition. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be slightly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
10. Tobacco smoking history of 10 pack years or greater, or ≥ 20 pack years if smoking cessation occurred at least 1 year prior to enrollment
11. Current use of antineoplastic drugs for other malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
To assess the disease control of participants who receive dose and volume-de-escalated radiotherapy to the neck, guided by treatment response through circulating tumor-modified HPV DNA testing | up to 2 years after radiotherapy
  Incidence of disease free survival as measured by circulating HPV on Nav Dx blood tests.

SECONDARY OUTCOMES:
To assess safety for treatment with reduced dose and volume-de-escalated radiotherapy to the neck | Evaluated through 6 months and 1 year post- radiation.
  Incidence of grade 3 (or greater) adverse events as defined by the CTCAE v5.0
To estimate quality of life of participants who receive reduced dose and volume-de-escalated radiotherapy to the neck | up to 2 years after radiotherapy
  Quality of life as determined by the EORTC H&N35. Questions are scaled from 1-4 with 1 meaning the symptom/problem was not experienced and 4 meaning the symptom/problem was experienced at a high level.
To estimate quality of life of participants who receive reduced dose and volume-de-escalated radiotherapy to the neck | up to 2 years after radiotherapy
  Quality of life as determined by the EORTC QLQ-C30. Majority of questions are scaled from 1-4 with 1 meaning the symptom/problem was not experienced and 4 meaning the symptom/problem was experienced at a high level. Two questions are scaled from 1-7 with 1 meaning very poor (worse outcome) and 7 meaning excellent (best outcome).

OTHER OUTCOMES:
To estimate long-term survival for participants treated with dose and volume-de-escalated radiotherapy to the neck | up to 5 years after radiotherapy
  Overall survival
To estimate the relationship between baseline lymphocyte counts and disease progression outcomes. | up to 2 years after radiotherapy
  Baseline lymphocyte counts from CBC with Differential blood test
To estimate the relationship between baseline lymphocyte counts and disease progression | up to 2 years after radiotherapy
  Occurrence of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Chris McLaughlin, M.D., Principal Investigator — UVA
Locations (5):
- United States (5):
  - Miami Cancer Institute, Miami, Florida
  - University of Virginia, Charlottesville, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Bon Secours, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No